CLINICAL TRIAL: NCT02337452
Title: The Patient-Driven Self-Navigated Web-Based Family Outreach Program for Cancer Prevention in High-Risk Families
Brief Title: Web-Based Family Outreach Program for Cancer Prevention in High-Risk Families
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2014-0715; NCI-2020-00567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0715 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (family outreach program): Patients communicate with at-risk family members to share genetic test results and other relevant information, as well as to learn more about their disease via family outreach program website. At risk family members are then contacted by a study coordinator or genetic counselor for further follow up. At-risk relatives receive resources to facilitate understanding of their at-risk status and to facilitate predictive testing.
  Interventions: Other: Questionnaire Administration; Behavioral: Web Site

INTERVENTIONS:
Other: Questionnaire Administration — Ancillary studies
Behavioral: Web Site — Communicate via family outreach program website
  Other Names: Internet Website; Website; www-website

SUMMARY:
This trial develops a patient-driven self-navigated web-based family outreach program for cancer prevention in high-risk families. Creating the family outreach program may help to improve the way in which genetic test results are communicated within families and increase the number of at-risk relatives who become aware of their risks.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a secure, web-based program for family outreach in Clinical Cancer Genetics (CCG).

II. The long-term goals of this program are expected to include, but are not limited to the following:

IIa. To enable families with inherited cancer susceptibility and/or at increased familial risk of cancer to provide personal and family history of neoplasia through a convenient and self-directed program.

IIb. To enable communication of possible inherited cancer susceptibility with and among family members through the web-based portal.

IIc. To facilitate genetic testing, screening and prevention strategies in those at risk.

IId. Establish high-risk cohort for optional participation in research and clinical trials.

OUTLINE:

Patients communicate with at-risk family members to share genetic test results and other relevant information, as well as to learn more about their disease via family outreach program website. At risk family members are then contacted by a study coordinator or genetic counselor for further follow-up. At-risk relatives receive resources to facilitate understanding of their at-risk status and to facilitate predictive testing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been diagnosed with a hereditary cancer-causing mutation. Individuals may be identified through clinical testing as patients at MD Anderson or patients whose mutation was identified at an outside institution who contact the registry
* Individuals that have clinical suspicion for syndromic cancer susceptibility, but in whom mutational testing has been nondiagnostic (depending on condition in question, nondiagnostic testing may be as little as 10%, as in familial adenomatous polyposis [FAP], or as high as 70% in suspected hereditary diffuse gastric cancer or HDGC)
* At-risk family members of individuals with a cancer causing mutation or of individuals with nondiagnostic testing notwithstanding presence of likely syndromic cancer. Such patients will in most cases not be MD Anderson patients. Note: The enrollment, consenting, and evaluation process anticipates and addresses this.

Exclusion Criteria:

* Index patients who test negative for a cancer causing mutation, except for those agreeing to provide family history (FH) that is informative for at-risk individuals when no other source of such information is available
* Patients who are unwilling or are unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with genetic abnormalities and their families at MD Anderson Cancer Center in Houston, Texas
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2048-04-30 (Estimated); Study Completion 2048-04-30 (Estimated)

PRIMARY OUTCOMES:
Web-Based Family Outreach Registry | Continual assessment of data over participant's life time (target follow-up duration: 40 Years)
  Data analysis for core functions of the web-based Family Outreach Registry will generally be descriptive. Web-based program to improve the way in which genetic test results are communicated within families and to increase the number of at-risk relatives who become aware of their risks.

CONTACTS AND LOCATIONS:
Overall Officials: Selvi Thirumurthi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org